CLINICAL TRIAL: NCT04848194
Title: Pleiotropic Role of TRPV1 in Psoriasis Inflammation
Acronym: TRIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 29BRC21.0013
Record Dates: First submitted 2021-04-07; First posted 2021-04-19 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Inflammation; Skin; Psoriasis
Keywords: psoriasis; TRVP1
MeSH Terms: conditions — Dermatitis; Psoriasis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients (Other): All patients with psoriasis recruted by dermatological departement.
  Interventions: Procedure: skin biopsy and blood sampling

INTERVENTIONS:
Procedure: skin biopsy and blood sampling — * 4 skin biopsies outside the face under local anesthesia: 2 in damaged zone, 2 in non-damage zone.
  * A blood sample

SUMMARY:
Widely expressed in the sensory nerve endings of the skin, Transient Receptor Potential Vanilloid 1 (TRPV1) is a receptor that plays an important role in the perception of pain and pruritus but also in skin inflammation, primarily by inducing the local release of several neuropeptides.

Although the mechanisms by which TRPV1-sensitizing inflammatory mediators in damaged skin have received considerable attention, the role of TRPV1 in psoriasis has so far been little explored.

However, two studies have reported that ablation of sensory nerves expressing TRPV1 reduced psoriasiform skin inflammation, demonstrating the neuronal contribution to inflammation in psoriasis.

However, the expression of TRPV1 is not limited to neurons alone. TRPV1 is also expressed by epidermal keratinocytes and skin microvessels.

For example, in 2018, transcriptomic analysis of psoriatic patient skins (by definition devoid of neuron nuclei) revealed that TRPV1 expression was increased in the skin of psoriatic patients suffering from itching (pruritus).

Regarding human keratinocytes, it is recognized that the activation of TRPV1 present on their surface induces the release of pro-inflammatory factors such as cyclooxygenase-2. In addition, the investigators have demonstrated that TRPV1 has a pivotal role in the keratinocyte production of inflammatory mediators, which is mediated by the protease-activated receptor-2 (PAR-2). However, the role of vascular TRPV1 in inflammation is not described.

The investigators hypothesize that in addition to neuronal TRPV1, non-neuronal TRPV1 receptors of non-neuronal cells (keratinocytes and endothelial cells) may be involved in the vicious circle of the inflammatory process characteristic of psoriasis. Putting TRPV1 at the center of the deregulation of the homeostatic balance including epithelial, neuronal and vascular inflammation in psoriasis is totally innovative.

DETAILED DESCRIPTION:
Each patient will have a sample taken in the dermatology department:

* 4 skin biopsies
* A blood sample.

Patients with psoriasis will be recruited from the dermatology department. There will be no further visits, so the duration of the study is 1 day.

The samples taken will be used to determine the pleiotropic role of TRPV1 in Psoriasis Inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old with psoriasis, with or without itching (pruritus).
* Presence of lesional and non lesional zones, in unexposed areas and surface area (outside the face and folds) large enough to allow the biopsies to be performed
* Patients who have given written consent

Exclusion Criteria:

* Patients with physical or psychological incapacity to sign consent
* Patients not covered by the Social Security system
* Patients with topical treatments for psoriasis,
* Patients with systemic treatments for psoriasis,
* Patients allergic to lidocaine
* Patients over the age of majority who are subject to legal protection or who are unable to give consent
* Patients deprived of liberty by a judicial or administrative decision
* Pregnant women, parturients and breastfeeding mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Role of TRPV1 receptors expressed by sensory neurons and non-neuronal cells (keratinocytes and endothelial cells) in the inflammatory process characteristic of psoriasis. | 1 day
  Density of intra-epidermal nerve fibers expressing the TRPV1 receptor

SECONDARY OUTCOMES:
Density changes of intra-epidermal nerve fibers expressing neuropeptides | 1 day
  Density of intra-epidermal nerve fibers expressing neuropeptides by immunohistochemistry
Changes in endothelial cell density between an injured and an uninjured area of the same patient | 1 day
  quantification of the transcriptional and protein expression of TRPV1
Changes in endothelial cell density between an injured and an uninjured area of the same patient | 1 day
  quantification of TRPV1 activity
Changes in endothelial cell density between an injured and an uninjured area of the same patient | 1 day
  Identification and quantification of the blood cytokine profile
Changes in the density of keratinocytes and their contacts with nerve fibers | 1 day
  Number and distribution of contacts between keratinocytes and nerve fibers

CONTACTS AND LOCATIONS:
Locations (1):
- TALAGAS, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.